CLINICAL TRIAL: NCT07391462
Title: Supporting Preventive Practices in Nutrition, Physical Activity and Sedentary Lifestyle in Primary Care: Amplifying the Potential of Opportunistic Interventions in Routine Consultations
Brief Title: Supporting Preventive Practices in Primary Care: Amplifying the Potential of Opportunistic Interventions
Acronym: APPRENDRE
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL21_1050; 24-5409 (Other: HCL)
Record Dates: First submitted 2026-01-29; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Sedentary; Suboptimal Health Status
Keywords: primary care; health behaviours; behaviour change techniques; co-construction; implementation science
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Brief opportunistic health behaviour change support group: Patients will receive a brief opportunistic behaviour change support on diet, physical activity and/or sedentary time by their trained General Practitioner (GP) during a routine consultation.
  Interventions: Behavioral: Training for GPs to learn healthy conversation skills for supporting patients' health behavior change
- Control group: Patients will be managed as usual during a routine consultation with their GP, without any special intervention.
  Interventions: Other: No training for GP

INTERVENTIONS:
Behavioral: Training for GPs to learn healthy conversation skills for supporting patients' health behavior change — GP training to deliver a brief opportunistic, behaviour change support on diet, physical activity and/or sedentary time to patients consulting them in routine practice.
  GPs in the intervention group will receive initial training (MOOC, C-MOOC and simulation workshops), follow-up training (feedback and personalized coaching), and toolkit of supporting materials for patients. Training and toolkit for GPs will be derived from Making Every Contact Counts materials and Cards for Change adapted to the French context and will be co-constructed with GP and patients.
  Groups: Brief opportunistic health behaviour change support group
Other: No training for GP — GP do not receive dedicated training for delivery of brief opportunistic behaviour change support to patients on diet, physical activity and/or sedentary time.
  Groups: Control group

SUMMARY:
In France, as worldwide, the prevalence of chronic conditions is increasing, with high burden on populations and healthcare systems. Behaviour is a key risk factor, and needs to be tackled within the social and environmental context in which it occurs. For example in 2017, the French eat too much processed food and salt, not enough fibers, 34% are overweight and 17% obese, and 80% present excessive sedentary time. In parallel, in France 5.4% of all cancers were attributable to sub-optimal nutrition (especially low fruits consumption and dietary fibers, and high processed meats consumption), and 6.3% to overweight/obesity or insufficient physical activity. Governments and health systems, including in France, have therefore considered a priority to intervene preventively on health behaviours throughout the lifespan.

For a populational approach to prevention via behaviour change, primary care professionals are best placed to intervene, due to the long-term relationship that can be established with healthcare users in their everyday life environments, and the many opportunities for brief interventions which can be delivered and followed up depending on individual needs. Research suggests that brief interventions can be effective in producing small but important changes in behaviour (Keyworth 2020) particularly if the intervention is based on a theoretical model of behaviour change (e.g., Prochaska's transtheoretical model or Bandura's cognitive social theory).

One such Public Health program is Making Every Contact Count (MECC), a program developed in England and deployed since 2007 and more recently implemented in Wales and Ireland as well. The development and implementation have been supported by epidemiological, behaviour change and implementation science research and continues to adapt to current challenges in preventive healthcare needs and provision. The "Healthy Conversation Skills" is a training program for healthcare professionals within the MECC program that focuses on how they can assess and support their patients' goals to improve behaviours such as physical activity and diet. It has been delivered since 2015 and shown effective (Adam 2020).

In France, 98% of general practitioners (GPs) consider prevention as part of their professional roles. However, initial and continuous training for primary care professionals focuses mainly on healthcare rather than prevention, and the latter is only addressed through physiological and epidemiological perspective but not on behaviour determinants and change techniques. Actually, there is at the moment limited training on assessing and supporting health behaviour change in primary care professionals in France, which limits the opportunities and effectiveness of a preventive approach to behavioural risk factors in chronic conditions. However, a direct transfer of the "Healthy Conversation Skills" program to the French context is unlikely to achieve optimal benefit, as differences in culture and health system organisation are considerable in behavioural care (de Bruin 2018). Collaborative approaches to developing and implementing training programs are recommended. The investigators therefore propose to co-construct a training program tailored to the context of GP practice in France, and study its effectiveness and implementation in supporting changes in diet, physical activity and sedentary time in adult patients from the general population consulting in routine care.

ELIGIBILITY:
Patients Inclusion Criteria:

* Age ≥ 18 years old
* Registered with a participating practice/practitioner
* Score < 5 for the "Stages of Change of Exercise Behaviour Scale" (pre-contemplation or contemplation stage) and/or Stage precontemplation or contemplation for the "Stages of Change for Healthy Diet Scale" (Precontemplation = answer to question 1 < 5 and answer to question 3 is no and Contemplation = answer to question 1 < 5, answer to question 3 is yes, and answer to question 4 is no).

Primary care professionals:

* GPs practicing in the Rhône-Alpes region
* Working in ambulatory care

Patients Exclusion Criteria:

* Being under guardianship and curatorship
* Pathological disordered eating (e.g., anorexia nervosa, bulimia nervosa,...)
* Acute severe pathology, life threatening condition
* Engaged in another research on diet or physical activity

Primary care professionals:

- Exclusive specialist practice (e.g., only sonography, angiology, addictiology , cosmetic surgery…)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target populations will be :
  * the general population aged 18 or over with sub-optimal health behaviours in terms of sedentary time or physical activity and diet, consulting in the practice of a GP recruited for the study for a routine consultation
  * GPs benefiting or not from the training evaluated
Sampling Method: Non-Probability Sample
Enrollment: 882 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Motivation for patients to change diet and/or physical activity behaviours, operationalsed as Readiness to change, measured by the "Stages of Change of Exercise Behaviour Scale" and the "Revised Dietary Stages of Change Measure" | At 2 weeks after the consultation
  Both scales measure motivation to practice regular physical activity or to increase daily portions of fruits and vegetables on a five-step scale corresponding to the stage of behavior change, according to the Prochaska's model.
  The primary endpoint will be considered as positive when reported score of at least one health behaviour is improved of at least one stage, compared to the pre-consultation score.
  The proportion of patients with improvement of at least one stage for at least one health behaviour will be analysed and compared between the two groups with a mixed logistic regression model.

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Dr Rémy BOUSSAGEON, Beynost
  - MSP D'Oullins, Oullins
  - MSP du 8 mai 1945, Saint-Priest
  - MSP Clos Caroline, Villeurbanne

IPD SHARING:
Plan to Share IPD: Undecided